CLINICAL TRIAL: NCT04805801
Title: Observational Study on the Safety of Hemlibra Subcutaneous Injection in Korean Hemophilia A Patients With/Without FVIII Inhibitors
Brief Title: The Safety of Emicizumab SC Injection in Korean Hemophilia A Patients With/Without FVIII Inhibitors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: JWP-HEM-401
Record Dates: First submitted 2021-03-17; First posted 2021-03-18 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Hemophilia A With Inhibitor; Hemophilia A Without Inhibitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Emicizumab Concentration Factor FVIII Inhibitor FVIII Activity
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemophilia A with FVIII inhibitors: Hemophilia A patients with FVIII inhibitors will administer Emicizumab at a loading dose of 3 mg/kg/week SC for the first 4 weeks of treatment followed by 1.5 mg/kg QW SC or 3mg/kg Q2W or 6mg/kg Q4W
  Interventions: Drug: Emicizumab subcutaneous injection
- Hemophilia A without FVIII inhibitors: Hemophilia A patients without FVIII inhibitors will administer Emicizumab at a loading dose of 3 mg/kg/week SC for the first 4 weeks of treatment followed by 1.5 mg/kg QW SC or 3mg/kg Q2W or 6mg/kg Q4W
  Interventions: Drug: Emicizumab subcutaneous injection

INTERVENTIONS:
Drug: Emicizumab subcutaneous injection — Safety and efficacy and PK, FVIII inhibitor titers will be evaluated by follow-up observation.
  Other Names: Emicizumab concentration, FVIII inhibitor titer, FVIII Activity lab test

SUMMARY:
To evaluate Safety and efficacy and pharmacokinetics, FVIII Inhibitor titers of Hemlibra subcutaneous injection (SC inj.) in Korean Hemophilia A patients with/without FVIII Inhibitors.

DETAILED DESCRIPTION:
Target subject :

1. Patients with Hemophilia A with FVIII inhibitors
2. Patients with severe Hemophilia A without FVIII inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Hemophilia A (congenital factor VIII deficiency) who will receive Hemlibra SC inj. according to medical decision by investigator
2. Signed informed consent form

Exclusion Criteria:

1. Subjects who are hypersensitive to Emicizumab
2. Subjects who are hypersensitive to mouse or hamster protein
3. Subjects with myocardial infarction or the history who are prohibited from administering L-Arginine containing drug
4. Subjects who participated in other clinical trials within a month before enrollment (or the first administration of Hemlibra SC inj.) (Unable to participate in other clinical trials related to Hemophilia A treatment even after enrollment)
5. Subjects who the investigator deems inappropriate for the study.
6. Moderate/Mild for Hemophilia A patients without FVIII inhibitors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1 .Hemophilia A patients with FVIII inhibitors 2. Severe Hemophilia A patients without FVIII inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2019-08-28 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Adverse events | for 24weeks
  AEs will be described for AEs and Adverse Drug Reactions (ADRs), Adverse Events of Special Interest (AESIs), other important AEs. Severity, outcome, causal relationship with study drug, etc. of AEs will be analyzed.

SECONDARY OUTCOMES:
Annualized Bleeding episode Rate (ABR) | for 24weeks
  The number of bleeds will be also annualized for each patient using the following formula

CONTACTS AND LOCATIONS:
Overall Officials: Chuhl Joo Lyu, Prof, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Severance Hospital, Seoul, South Korea